CLINICAL TRIAL: NCT03847012
Title: The Blood Pressure Responses to Different Exercise Models in Patients With Coronary Artery Disease
Brief Title: Blood Pressure Responses to Different Exercise Modes in Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201807117RIND
Record Dates: First submitted 2019-02-10; First posted 2019-02-20 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; blood pressure; rehabilitation; exercise mode
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with coronary artery diseases (Experimental): The investigators will recruit 30 subjects with CAD who are referred to phase II cardiopulmonary rehabilitation exercise training. After at least 3 times of familiar with the cardiopulmonary rehabilitation training machine, the subjects performed the treadmill or stationary bicycle and exercise to personalized target heart rate for 10 minutes, take a rest until the heart rate recover to the resting heart rate, and then repeated the exercise in another exercise mode.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — The test order will be random. After at least 12 times of cardiopulmonary rehabilitation training, the test will be performed again.

SUMMARY:
The purposes of this study were to compare blood pressure responses of the same target heart rate on different exercise modes in patients with coronary artery diseases (CAD) and to compare the effects of blood pressure responses after exercise training.

The investigators will recruit 30 subjects with CAD who are referred to phase II cardiopulmonary rehabilitation exercise training. The subjects performed the treadmill or stationary bicycle exercise randomly.

DETAILED DESCRIPTION:
Considering cardiopulmonary rehabilitation intensity is often setting by heart rate clinically, and only few study focused on exercise responses patients with CAD, the purposes of this study were to compare blood pressure responses of the same target heart rate on different exercise modes in patients with CAD and to compare the effects of blood pressure responses after exercise training.

This is a crossover trial study. The investigators will recruit 30 subjects with CAD who are referred to phase II cardiopulmonary rehabilitation exercise training. After at least 3 times of familiar with the cardiopulmonary rehabilitation training machine, the subjects performed the treadmill or stationary bicycle and exercise to personalized target heart rate for 10 minutes, take a rest until the heart rate recover to the resting heart rate, and then repeated the exercise in another exercise mode. The test order will be random. After at least 12 times of cardiopulmonary rehabilitation training, the test will be performed again.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery diseases who are referred to phase II cardiopulmonary rehabilitation exercise training.

Exclusion Criteria:

* patients with non-coronary artery diseases
* atrial fibrillation
* neurological or musculoskeletal problems

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
heart rate | Change from baseline heart rate at 6 weeks
  heart rate
blood pressure | Change from baseline blood pressure at 6 weeks
  blood pressure

SECONDARY OUTCOMES:
perceived exertion scale | baseline and 6 weeks
  how effort the participant feel. Range from 1to 10. Higher values represent harder.
heart rate variability | baseline and 6 weeks
  heart rate variability

OTHER OUTCOMES:
age | baseline
  questionnaire
gender | baseline
  questionnaire
risk level of exercise | baseline
  AACVPR Stratification Algorithm for Risk of Event. Include high, moderate and low risk
co-morbidity | baseline
  questionnaire
medication | baseline
  questionnaire
level of exercise intensity | baseline
  percent of heart rate reserve

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No